CLINICAL TRIAL: NCT00490646
Title: Randomized Phase II Study of Ixabepilone Plus Trastuzumab vs. Docetaxel Plus Trastuzumab in Female Subjects With Her2+ Locally Advanced and/or Metastatic Breast Cancer
Brief Title: A Phase II Combination of Trastuzumab and Ixabepilone Versus Trastuzumab and Docetaxel in Patients With Advanced and/or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-140; Eudract No: 2007-000721-21
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
Keywords: Locally advanced and/or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Epothilones; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): trastuzumab 4 mg/kg loading dose, then 2 mg/kg weekly + ixabepilone 40 mg/m^2 intravenous (IV) over 3 hours once every 21 days (using a 21-day cycle); until disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone; Drug: trastuzumab
- Arm B (Active Comparator): trastuzumab 4 mg/kg loading dose, then 2 mg/kg weekly + docetaxel 100 mg/m^2 IV over 1 hour once every 21 days (using a 21-day cycle); until disease progression or unacceptable toxicity.
  Interventions: Drug: docetaxel; Drug: trastuzumab

INTERVENTIONS:
Drug: ixabepilone — Ixabepilone 40 mg/m^2 was administered as a 3-hour I.V. continuous infusion on Day 1 in a 21-day cycle until disease progression or unacceptable toxicity.
  For the first cycle, ixabepilone was administered the day following the first dose of trastuzumab (in the first cycle trastuzumab was given on Day 0); in all the following cycles, ixabepilone was administered immediately after the subsequent doses of trastuzumab if the preceding dose of trastuzumab was well tolerated.
  Other Names: BMS-247550; Epothilone; IXEMPRA®
  Arms: Arm A
Drug: docetaxel — Docetaxel 100 mg/m^2 was administered as a 1-hour IV continuous infusion on Day 1 in a 21-day cycle until disease progression or unacceptable toxicity. For the first cycle, docetaxel was administered the day following the first dose of trastuzumab (i.e. in the first cycle trastuzumab was given on Day 0); in all following cycles, docetaxel was administered immediately after trastuzumab if the preceding dose of trastuzumab was well tolerated.
  Arms: Arm B
Drug: trastuzumab — Trastuzumab was administered as an IV infusion on Days 1, 8, and 15 of each 21-day cycle at a dose of 2 mg/kg until disease progression or unacceptable toxicity. In cycle 1, a loading dose of 4 mg/kg was administered as a 90-minute IV infusion on a day before initial administration of chemotherapy (i.e. on Day 0). Trastuzumab was given immediately prior to ixabepilone (Arm A) or docetaxel (Arm B) in all subsequent cycles as a 30-minute IV infusion if the initial dose was well tolerated.

SUMMARY:
The purpose of this randomized, Phase 2 open-label study was to assess the response rate of participants with Human Epidermal Growth Factor Receptor 2 (Her2+) locally advanced and/or metastatic breast cancer (not previously treated with chemotherapy or trastuzumab) to treatment with ixabepilone plus trastuzumab and/or docetaxel plus trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic HER2+ breast cancer not previously treated with chemotherapy or trastuzumab.
* Subjects who had received prior (neo)adjuvant chemotherapy or trastuzumab were eligible except if they relapsed within 12 months after the last dose of a taxane or trastuzumab given as (neo)adjuvant therapy.
* Measurable disease
* Left Ventricular Ejection Fraction (LVEF) ≥50%

Exclusion Criteria:

* Prior chemotherapy or trastuzumab for metastatic breast cancer (MBC)
* Relapse within 1 year after (neo)adjuvant taxane or trastuzumab
* Neuropathy > Grade 1
* Significant cardiovascular disease
* Any brain metastases

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- France (4):
  - Local Institution, Caen
  - Local Institution, Grenoble
  - Local Institution, Saint-Priest-en-Jarez
  - Local Institution, Toulouse
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Pireaus
- Italy (6):
  - Local Institution, Bologna
  - Local Institution, Brescia
  - Local Institution, Modena
  - Local Institution, Napoli
  - Local Institution, Roma
  - Local Institution, Sora
- Local Institution, Madrid, Spain
- Turkey (Türkiye) (2):
  - Local Institution, Ankara
  - Local Institution, Izmir

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV: trastuzumab 4 mg/kg loading dose, then 2 mg/kg weekly + ixabepilone 40 mg/m^2 intravenous (IV) over 3 hours once every 21 days (using a 21-day cycle); until disease progression or unacceptable toxicity.
- Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV: trastuzumab 4 mg/kg loading dose, then 2 mg/kg weekly + docetaxel 100 mg/m^2 IV over 1 hour once every 21 days (using a 21-day cycle); until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Started | 25 | 25
Treated | 24 | 24
Completed | 23 (Completed=Off-treatment (Major reasons: Disease progression=14; study drug toxicity=4)) | 23 (Completed=Off-treatment (Major reasons: Disease progression=13; study drug toxicity=1))
Not Completed | 2 | 2
Not completed — Still on trastuzumab monotherapy | 1 | 1
Not completed — Never Treated (had an adverse event) | 1 | 0
Not completed — Never Treated (withdrew consent) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Median (Full Range); unit: years] | 52.0 [29.0 to 71.0] | 53.0 [37.0 to 82.0] | 52.5 [29.0 to 82.0]
Age, Customized [Number; unit: participants]
  < 65 years | 19 | 21 | 40
  >=65 years | 6 | 4 | 10
Sex/Gender, Customized [Number; unit: participants]
  Female | 25 | 25 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 25 | 50
Karnofsky Performance Status [Number; unit: participants] — Karnofsky Performance Status classifies participants according to their functional impairment. Scores range from 0-100 units on a scale; lower the score, the worse the survival for most serious illnesses.
  100: Normal, no complaints. 90: Able to carry on normal activities; minor signs or symptoms of disease. 80: Normal activity with effort. 70: Cares for self. Unable to carry on normal activity or to do active work. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Scores were converted to Karnofsky Performance Status Scores.
  participants
    100 | 15 | 15 | 30
    90 | 5 | 9 | 14
    80 | 4 | 0 | 4
    70 | 1 | 0 | 1
    Not Reported | 0 | 1 | 1
Menopausal Status [Number; unit: participants]
  Pre-menopausal | 8 | 6 | 14
  Peri-menopausal | 1 | 2 | 3
  Post-menopausal | 14 | 15 | 29
  Not Reported | 2 | 2 | 4
Number of participants who received prior chemotherapy in neoadjuvant/adjuvant setting [Number; unit: participants] | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR; Assessed by Response Evaluation Criteria in Solid Tumors [RECIST] Version 1.1)
Description: Percentage of participants with best overall response (BOR) of either complete response (CR) or partial response (PR) according to RECIST version 1.1 as determined by the investigator. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (LD) of all lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. A two-sided confidence interval (CI) was computed using the Clopper-Pearson method.
Time Frame: Assessed every 6 weeks from initiation of study therapy up to 12 months; then every 3 months until disease progression (maximum time that any participant was on therapy was 108 weeks)
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 25 | 25
percentage of participants | 60.0 [38.7 to 78.9] | 52.0 [31.3 to 72.2]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in months from randomization until first date of documented progressive disease (PD) or death from any cause without prior documentation of progression. PD=≥20% increase in sum of LD of target lesions in reference to smallest sum LD recorded at or following baseline or unequivocal progression of existing non-target lesion(s) overall.
  Estimated by the Kaplan-Meier product limit method. A two-sided 95% CI for median duration was computed by the Brookmeyer and Crowley method.
Time Frame: From randomization until the first date of documented progressive disease (PD) or death from any cause without prior documentation of progression (maximum participant PFS of 39.7 months).
Population: All randomized participants. Participants who did not progress or died were censored on the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 25 | 25
months | 11.3 [5.8 to 16.8] | 13.0 [6.7 to 21.6]

3. Secondary Outcome: Time to Response
Description: Time to response was defined as the time in weeks from randomization until the measurement criteria are first met for a CR or PR, whichever is recorded first.
  CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the LD of all lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. Estimated by the Kaplan-Meier product limit method. A two-sided 95% CI for median duration was computed by the Brookmeyer and Crowley method.
Time Frame: From randomization every 6 weeks for first 12 months and thereafter every 3 months until CR or PR whichever was recorded first (maximum participant time to response of 18.4 weeks.)
Population: All randomized participants with CR or PR.
Measure: Median (Full Range); unit: weeks
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 15 | 13
weeks | 10.1 [5.9 to 18.4] | 7.3 [5.0 to 18.1]

4. Secondary Outcome: Duration of Response
Description: Period measured in months from time that measurement criteria were first met for CR or PR until first date of documented PD or death from any cause without prior documentation of progression.
  PD=≥20% increase in sum of LD of target lesions in reference to smallest sum LD recorded at or following baseline or unequivocal progression of existing non-target lesion(s) overall. Refer to Outcome Measure 1 for definitions of CR and PR. Estimated by the Kaplan-Meier product limit method. A two-sided 95% CI for median duration was computed by Brookmeyer and Crowley method.
Time Frame: From the date of first PR or CR assessment to the date of documented progressive disease or death without prior documentation of progression (maximum participant duration of response of 38 months.)
Population: All randomized participants with CR or PR. The participants who neither relapsed nor died were censored on the date of their last tumor assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 15 | 13
months | 11.5 [6.8 to 21.4] | 16.5 [7.2 to NA] — Data insufficient to estimate the upper limit of the confidence interval.

5. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Adverse Events (AEs), and AEs Leading to Discontinuation of Study Therapy Per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 3.0
Description: AE: New untoward medical occurrence or worsening of a preexisting medical condition that does not have causal relationship with this treatment. SAE: Untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, drug dependency/abuse; life-threatening, an important medical event, a congenital anomaly/birth defect; requires inpatient hospitalization/prolongs existing hospitalization. Grade 3=Severe; and Grade 4=Life-threatening or disabling. GR=Grade.
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug (maximum time that any participant was on therapy was 108 weeks.)
Population: Treated participants: Participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 24 | 24
participants
  All deaths | 1 | 1
  Death within 30 days of last dose of study therapy | 1 | 0
  SAEs (Any Grade) | 6 | 13
  SAEs (Grades 3-4) | 4 | 12
  Drug-related SAEs (Any Grade) | 3 | 10
  Drug-related SAEs (Grades 3-4) | 2 | 8
  AEs (Any Grade) | 24 | 24
  AEs (Grades 3-4) | 19 | 23
  Drug-related AEs (Any Grade) | 24 | 24
  Drug-related AEs (Grades 3-4) | 18 | 22
  AEs leading to discontinuation of therapy (Any GR) | 5 | 9
  AEs leading to discontinuation of therapy (GR 3-4) | 2 | 4
  Drug-related peripheral neuropathy (Any Grade) | 16 | 12
  Drug-related peripheral neuropathy (Grades 3-4) | 2 | 0

6. Secondary Outcome: Number of Participants With Hematology Abnormalities by Worst Grade Per National Cancer Institute Common Terminology Criteria Adverse Events (NCI CTCAE), Version 3.0
Description: Grade (GR)1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. White blood cell (WBC):GR1=<LLN-3.0*10^9/L; GR2=<3.0-2.0*10^9/L; GR3=<2.0-1.0*10^9/L; GR4=<1.0*10^9/L. Absolute Neutrophil Count (ANC):GR1=<LLN-1.5*10^9 /L; GR2=<1.5-1.0*10^9/L; GR3=<1.0-0.5*10^9/L; GR4=<0.5*10^9/L. Platelets:GR1=<LLN-75.0*10^9/L; GR2=<75.0-50.0*10^9/L; GR3=<50.0-25.0*10^9/L, GR4=<25.0*10^9/L. Hemoglobin:GR1=<LLN-10.0g/dL; GR2=<10.0-8.0g/dL; GR3=<8.0-6.5g/dL, GR4=<6.5g/dL. LLN=lower limit of normal.
Time Frame: Prior to every cycle of therapy (i.e. before starting of every 21 day or 3 week cycle; maximum time that any participant was on therapy was 108 weeks.)
Population: Treated participants: Participants who received at least 1 dose of study therapy. n=number of participants with measures available.
Measure: Number; unit: participants
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 24 | 24
participants
  WBC Grade 1 (n=24; n=22) | 6 | 1
  WBC Grade 2 (n=24; n=22) | 7 | 1
  WBC Grade 3 (n=24; n=22) | 8 | 15
  WBC Grade 4 (n=24; n=22) | 1 | 4
  ANC Grade 1 (n=23; n=23) | 2 | 0
  ANC Grade 2 (n=23; n=23) | 4 | 0
  ANC Grade 3 (n=23; n=23) | 8 | 3
  ANC Grade 4 (n=23; n=23) | 6 | 19
  Platelet Count Grade 1 (n=24; n=23) | 9 | 3
  Platelet Count Grade 2 (n=24; n=23) | 0 | 0
  Platelet Count Grade 3 (n=24; n=23) | 0 | 0
  Platelet Count Grade 4 (n=24; n=23) | 1 | 0
  Hemoglobin Grade 1 (n=24; n=23) | 14 | 12
  Hemoglobin Grade 2 (n=24; n=23) | 8 | 8
  Hemoglobin Grade 3 (n=24; n=23) | 0 | 1
  Hemoglobin Grade 4 (n=24; n=23) | 0 | 0

7. Secondary Outcome: Number of Participants With Serum Chemistry Abnormalities by Worst Grade Per National Cancer Institure Common Terminology Criteria Adverse Events (NCI CTCAE), Version 3.0
Description: Grading: NCI CTCAE, Version 3.0. GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening or disabling. Normal ranges provided by local laboratory and may also vary by age and sex. Alkaline phosphatase (ALP), alanine aminotransferase (ALT), and aspartate aminotransferase (AST): GR1=>ULN-2.5*ULN; GR2=>2.5-5.0*ULN; GR3=>5.0-20.0*ULN; GR4=>20.0*ULN. Total bilirubin: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3-10*ULN, GR4=>10*ULN. Creatinine: GR1=>ULN-1.5*ULN, GR2=>1.5-3.0*ULN, GR3=>3.0-6.0*ULN, GR4=>6.0*ULN. ULN=upper limit of normal.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 24 | 24
participants
  ALP Grade 1 (n=23; n=23) | 11 | 8
  ALP Grade 2 (n=23; n=23) | 0 | 1
  ALP Grade 3 (n=23; n=23) | 0 | 0
  ALP Grade 4 (n=23; n=23) | 0 | 0
  ALT Grade 1 (n=24; n=23) | 10 | 15
  ALT Grade 2 (n=24; n=23) | 3 | 0
  ALT Grade 3 (n=24; n=23) | 0 | 1
  ALT Grade 4 (n=24; n=23) | 0 | 0
  AST Grade 1 (n=24; n=23) | 13 | 11
  AST Grade 2 (n=24; n=23) | 0 | 1
  AST Grade 3 (n=24; n=23) | 1 | 0
  AST Grade 4 (n=24; n=23) | 0 | 0
  Total Bilirubin Grade 1 (n=24; n=23) | 2 | 2
  Total Bilirubin Grade 2 (n=24; n=23) | 0 | 0
  Total Bilirubin Grade 3 (n=24; n=23) | 1 | 0
  Total Bilirubin Grade 4 (n=24; n=23) | 0 | 0
  Creatinine Grade 1 (n=24; n=23) | 2 | 1
  Creatinine Grade 2 (n=24; n=23) | 2 | 0
  Creatinine Grade 3 (n=24; n=23) | 0 | 0
  Creatinine Grade 4 (n=24; n=23) | 0 | 0

8. Primary Outcome: Number of Participants With Best Overall Response (BOR) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: BOR was the best response recorded from the start of treatment until disease progression or recurrence (taking the smallest measurement recorded since the start of treatment as reference). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the LD of all lesions. CR and PR criteria should be met again after 4 weeks and before 6 weeks after initial assessment. Stable disease (SD)=Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. Refer to Outcome Measure 3 for definition of PD.
Time Frame: as for outcome 1
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV
Number analyzed (Participants) | 25 | 25
participants
  Complete response | 3 | 2
  Partial response | 12 | 11
  Stable disease | 6 | 9
  Progressive disease | 1 | 1
  Unable to determine (UTD; Death due to toxicity) | 1 | 0
  UTD (reason other than toxicity or progression) | 1 | 1
  Never treated | 1 | 1

ADVERSE EVENTS:
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug (maximum time that any participant was on therapy was 108 weeks.)
Arm/Group | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV
Serious Adverse Events (participants affected / at risk) | 13/24 | 6/24
Other Adverse Events (participants affected / at risk) | 23/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV (N=24) | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV (N=24)
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
ATAXIA (Nervous system disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 0
HAEMATOTOXICITY (Blood and lymphatic system disorders) | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
APLASIA (Congenital, familial and genetic disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
EXTRAVASATION (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab 2 mg/kg + Docetaxel 100 mg/m^2 IV (N=24) | Trastuzumab 2 mg/kg + Ixabepilone 40 mg/m^2 IV (N=24)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 5
NEUTROPHIL COUNT (Investigations) | 1 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 1
CONSTIPATION (Gastrointestinal disorders) | 3 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 5
PALPITATIONS (Cardiac disorders) | 0 | 2
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 0
STOMATITIS (Gastrointestinal disorders) | 4 | 2
WEIGHT INCREASED (Investigations) | 3 | 4
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 | 6
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 2
LACRIMATION INCREASED (Eye disorders) | 2 | 0
MUCOSAL INFLAMMATION (General disorders) | 6 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 4 | 3
PARAESTHESIA (Nervous system disorders) | 4 | 8
PYREXIA (General disorders) | 9 | 4
VOMITING (Gastrointestinal disorders) | 4 | 5
ASTHENIA (General disorders) | 5 | 8
DERMATITIS (Skin and subcutaneous tissue disorders) | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 2 | 2
NEUROTOXICITY (Nervous system disorders) | 1 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 | 3
ANAEMIA (Blood and lymphatic system disorders) | 8 | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 | 2
DIARRHOEA (Gastrointestinal disorders) | 12 | 7
DIZZINESS (Nervous system disorders) | 0 | 2
FATIGUE (General disorders) | 5 | 4
HAEMOGLOBIN DECREASED (Investigations) | 1 | 2
HYPERSENSITIVITY (Immune system disorders) | 2 | 5
HYPERTENSION (Vascular disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 14 | 11
PHARYNGITIS (Infections and infestations) | 1 | 4
SENSORY LOSS (Nervous system disorders) | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 3
INFLUENZA LIKE ILLNESS (General disorders) | 2 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 4
NEUTROPHIL COUNT DECREASED (Investigations) | 4 | 3
PAIN (General disorders) | 2 | 5
ALOPECIA (Skin and subcutaneous tissue disorders) | 7 | 9
DEPRESSION (Psychiatric disorders) | 0 | 3
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 3
HEADACHE (Nervous system disorders) | 2 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 8
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3
INSOMNIA (Psychiatric disorders) | 1 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 6
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 2
OEDEMA PERIPHERAL (General disorders) | 4 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 7 | 7
TACHYCARDIA (Cardiac disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.